CLINICAL TRIAL: NCT04986618
Title: Investigation of the Effects of One-Way and Two-Way Nordic Exercise on the Agility of Active Children
Brief Title: The Effect of Nordic Exercise on Children's Agility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Murat EMİRZEOĞLU, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-38
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Sports Performance in Children
Keywords: soccer; child; agility; nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One-way Nordic Exercise Group (Experimental)
  Interventions: Other: One-way Nordic Exercise
- Two-way Nordic Exercise Group (Experimental)
  Interventions: Other: Two-way Nordic Exercise
- Control Group (No Intervention)

INTERVENTIONS:
Other: One-way Nordic Exercise — Participants in this group will be given the standard Nordic Hamstring exercise.
  Arms: One-way Nordic Exercise Group
Other: Two-way Nordic Exercise — In addition to the standard Nordic Hamstring exercise, participants in this group will do the same exercise backwards for the quadriceps.
  Arms: Two-way Nordic Exercise Group

SUMMARY:
The aim of this research is to investigate the effect of one-way and two-way Nordic exercise on the agility of active children. Children who meet the necessary criteria will be randomly assigned to one-way Nordic exercise group, two-way Nordic exercise group and control group by drawing lots. Volunteers in the training group will participate in a four-week training, two sessions per week. Agility will be assessed at baseline and after four weeks with the T-agility test. In-group and between-group comparisons will be analyzed using the Statistical Package for the Social Sciences program and appropriate tests.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 8-12
* To be actively participating in football training.

Exclusion Criteria:

* Those with orthopedic, neurological and congenital problems.
* Those with any systematic disease.
* Those who have experience taping before.
* Those who have undergone any surgery within the last 1 year.
* Those who have been absent from training for more than 2 weeks in the last three months.

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
T-Agility Test | 4 week
  Agility

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)